CLINICAL TRIAL: NCT00143468
Title: The Specific Elastance in Acute Lung Injury/Acute Respiratory Distress Syndrome (ALI/ARDS) Patients: Barotrauma and Volutrauma
Brief Title: The Specific Elastance in Acute Lung Injury/Acute Respiratory Distress Syndrome (ALI/ARDS) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Policlinico Hospital (Other)
Responsible Party: Principal Investigator, Davide Chiumello, MD, Policlinico Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1160
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2011-12-01 (Estimated); Status verified 2011-11

CONDITIONS: Acute Lung Injury; ARDS
Keywords: gas exchange; respiratory mechanics
MeSH Terms: conditions — Acute Lung Injury | interventions — Respiration, Artificial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): ALI/ARDS patients and healthy subjects
  Interventions: Behavioral: mechanical ventilation

INTERVENTIONS:
Behavioral: mechanical ventilation — measurement of specific lung elastance during mechanical ventilation

SUMMARY:
The investigators aim to study the specific elastance in ALI/ARDS patients during invasive mechanical ventilation.

DETAILED DESCRIPTION:
In sedated and paralyzed ALI/ARDS patients, we studied the specific elastance and also, we compared the specific elastance to healthy subjects during invasive mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Stable ALI/ARDS patients during invasive mechanical ventilation

Exclusion Criteria:

* Hemodynamic failure, pneumothorax

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2005-03; Primary Completion 2007-03 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Specific elastance | 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: davide chiumello, MD, Principal Investigator — Policlinico Hospital
Locations (1):
- Ospedale policlinico, Milan, Milano, Italy

REFERENCES:
- [Derived] Chiumello D, Carlesso E, Cadringher P, Caironi P, Valenza F, Polli F, Tallarini F, Cozzi P, Cressoni M, Colombo A, Marini JJ, Gattinoni L. Lung stress and strain during mechanical ventilation for acute respiratory distress syndrome. Am J Respir Crit Care Med. 2008 Aug 15;178(4):346-55. doi: 10.1164/rccm.200710-1589OC. Epub 2008 May 1. PMID 18451319